CLINICAL TRIAL: NCT04544306
Title: Partial Oral Antimicrobial Versus Intravenous Antimicrobial Therapy to Treat Infective Endocarditis in People Who Inject Drugs
Brief Title: Partial Oral Antimicrobials to Treat Infective Endocarditis in People Who Inject Drugs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Silverman, MD, Chair/Chief,Infectious Diseases Division, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10418
Record Dates: First submitted 2020-08-25; First posted 2020-09-10 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Infective Endocarditis
Keywords: PWID; oral antibiotics; endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Standard of Care (intravenous antimicrobial therapy according to the American Heart Association Guideline 2015)
- Partial oral treatment arm (Experimental): The mode of antimicrobial delivery is switched to oral therapy after at least 10 days of IV therapy, guided by antimicrobial susceptibility
  Interventions: Other: Partial oral antimicrobial therapy

INTERVENTIONS:
Other: Partial oral antimicrobial therapy — Switch intravenous antimicrobial therapy to oral after an initial period of 10 days to oral antimicrobial therapy. Antimicrobial choices will be guided by antimicrobial susceptibilities.
  Arms: Partial oral treatment arm

SUMMARY:
Infective endocarditis (IE) is a serious infection associated with significant morbidity and mortality. Recent studies demonstrated an increased risk of infective endocarditis in people who inject drugs (PWIDs). PWIDs have a high rate of non-compliance with hospital admissions and leaving against medical advice. A recent landmark randomized controlled trial demonstrated similar outcomes when comparing partial oral antimicrobial therapy to continued intravenous antimicrobial therapy in the general population. Performing a trial to explore the non-inferiority of oral compared to intravenous antimicrobial therapy in PWIDs is essential in advancing patient care in this high risk increasing population.

DETAILED DESCRIPTION:
This is a randomized open-label study. Participants will be randomized 1:1 in blocks of 5 to either continued intravenous antimicrobial therapy or oral antimicrobial therapy after a minimum of 10 days of IV therapy. The antimicrobial choice will be based on antimicrobial susceptibility. All oral regimens for gram-positive organisms will include 2 different agents. Gram-negative pathogens will be treated with oral quinolones if susceptibility results are compatible. Decisions regarding ongoing inpatient or outpatient therapy will be made at the discretion of the attending physician. Outpatient follow up will be once weekly for 6 weeks and then at 3 months. At each follow-up visit, participants will undergo a general physical exam, and their adherence to therapy and general wellbeing will be assessed as well. Blood samples will be sent for a complete blood count, creatinine, C-reactive protein by the investigators to ensure continued improvement in response to therapy. Within 72 hours of stopping therapy, a transthoracic echocardiogram will be performed to determine response to therapy and to establish a new baseline to which subsequent echocardiograms if medically indicated would be compared to assess for relapse or development of a new IE. All lab tests are done at our affiliated hospitals. Investigators plan first on performing a feasibility study. In the feasibility study, investigators recruit a total of 50 patients and randomize 25 in each arm. Baseline characteristics, of clinical interest with a potential impact on prognosis, and patients' outcomes will be compared using the Chi-square test for categorical variables and the t-test and the Mann-Whitney test for continuous variables, when appropriate. To examine the association between oral antimicrobial therapy and 90-day mortality, investigators plan to perform a multivariable logistic regression analysis with oral therapy being the independent variable. The model will also include variables of clinical interest: diabetes, renal impairment, immune-compromising condition, age > 50, and evidence of embolization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years with self-reported intravenous drug use within 3 months of admission
2. Transthoracic and/or transesophageal echocardiogram for IE diagnosis should be done within 48 hours of randomization
3. Patients meet the modified Duke criteria for possible or definite infective endocarditis diagnosis
4. Infection with an organism susceptible to at least two oral antimicrobial agents from different classes. In gram-negative bacterial endocarditis, susceptibility to fluoroquinolones only would be acceptable for inclusion
5. Polymicrobial infections may be enrolled if an acceptable oral regimen can be constructed containing at least 2 agents against each gram-positive organism and one against each gram-negative
6. Fungal Endocarditis may be enrolled if susceptibility to an oral azole is confirmed
7. IE Patients who demonstrate improvement with initial intravenous therapy will be recruited
8. Patients should receive a minimum of 10 days initial IV therapy and should have a minimum of 14 days remaining of their antimicrobial therapy

Exclusion Criteria:

1. Undrained valvular, perivalvular, or cardiac abscess on echocardiogram studies
2. Failure to show improvement to initial intravenous antimicrobial therapy
3. Oral antibiotic malabsorption due to gastrointestinal disorders
4. Acutely intoxicated patients who are not able to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of eligible participants who are approached for consent to participate will be recorded. | 18 months
  Number of individuals who are eligible to be enrolled during the study time frame.
The percentage who consent for enrollment will be determined as well as the reasons for refusal. | 18 months
  Number of patients that participate as well as those who refuse to enroll during the study time frame.

SECONDARY OUTCOMES:
Percentage of enrolled patients for whom 90 day survival data is able to be confirmed. | 3 months after randomization
  Number of patients with all cause death or survival documented at 90 days post enrollment.
Percentage of enrolled patients who continue in their assigned treatment arm (Oral or Parenteral) throughout the treatment interval. | 6 weeks post enrollment
  The assessment of compliance with oral or parenteral antibiotics will be carried out during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, MD,FRCP, Principal Investigator — LHSC
Locations (2):
- Canada (2):
  - University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tookes H, Diaz C, Li H, Khalid R, Doblecki-Lewis S. A Cost Analysis of Hospitalizations for Infections Related to Injection Drug Use at a County Safety-Net Hospital in Miami, Florida. PLoS One. 2015 Jun 15;10(6):e0129360. doi: 10.1371/journal.pone.0129360. eCollection 2015. PMID 26075888
- [Background] Weir MA, Slater J, Jandoc R, Koivu S, Garg AX, Silverman M. The risk of infective endocarditis among people who inject drugs: a retrospective, population-based time series analysis. CMAJ. 2019 Jan 28;191(4):E93-E99. doi: 10.1503/cmaj.180694. PMID 30692105
- [Background] Iversen K, Ihlemann N, Gill SU, Madsen T, Elming H, Jensen KT, Bruun NE, Hofsten DE, Fursted K, Christensen JJ, Schultz M, Klein CF, Fosboll EL, Rosenvinge F, Schonheyder HC, Kober L, Torp-Pedersen C, Helweg-Larsen J, Tonder N, Moser C, Bundgaard H. Partial Oral versus Intravenous Antibiotic Treatment of Endocarditis. N Engl J Med. 2019 Jan 31;380(5):415-424. doi: 10.1056/NEJMoa1808312. Epub 2018 Aug 28. PMID 30152252
- [Background] Kasper KJ, Manoharan I, Hallam B, Coleman CE, Koivu SL, Weir MA, McCormick JK, Silverman MS. A controlled-release oral opioid supports S. aureus survival in injection drug preparation equipment and may increase bacteremia and endocarditis risk. PLoS One. 2019 Aug 9;14(8):e0219777. doi: 10.1371/journal.pone.0219777. eCollection 2019. PMID 31398210
- [Background] Rodger L, Glockler-Lauf SD, Shojaei E, Sherazi A, Hallam B, Koivu S, Gupta K, Hosseini-Moghaddam SM, Silverman M. Clinical Characteristics and Factors Associated With Mortality in First-Episode Infective Endocarditis Among Persons Who Inject Drugs. JAMA Netw Open. 2018 Nov 2;1(7):e185220. doi: 10.1001/jamanetworkopen.2018.5220. PMID 30646383
- [Background] Rodger L, Shah M, Shojaei E, Hosseini S, Koivu S, Silverman M. Recurrent Endocarditis in Persons Who Inject Drugs. Open Forum Infect Dis. 2019 Sep 9;6(10):ofz396. doi: 10.1093/ofid/ofz396. eCollection 2019 Oct. PMID 31660358
- [Background] Baddour LM, Wilson WR, Bayer AS, Fowler VG Jr, Tleyjeh IM, Rybak MJ, Barsic B, Lockhart PB, Gewitz MH, Levison ME, Bolger AF, Steckelberg JM, Baltimore RS, Fink AM, O'Gara P, Taubert KA; American Heart Association Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Stroke Council. Infective Endocarditis in Adults: Diagnosis, Antimicrobial Therapy, and Management of Complications: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2015 Oct 13;132(15):1435-86. doi: 10.1161/CIR.0000000000000296. Epub 2015 Sep 15. PMID 26373316
- [Background] Heldman AW, Hartert TV, Ray SC, Daoud EG, Kowalski TE, Pompili VJ, Sisson SD, Tidmore WC, vom Eigen KA, Goodman SN, Lietman PS, Petty BG, Flexner C. Oral antibiotic treatment of right-sided staphylococcal endocarditis in injection drug users: prospective randomized comparison with parenteral therapy. Am J Med. 1996 Jul;101(1):68-76. doi: 10.1016/s0002-9343(96)00070-8. PMID 8686718
- [Background] Al-Omari A, Cameron DW, Lee C, Corrales-Medina VF. Oral antibiotic therapy for the treatment of infective endocarditis: a systematic review. BMC Infect Dis. 2014 Mar 13;14:140. doi: 10.1186/1471-2334-14-140. PMID 24624933
- [Background] Tissot-Dupont H, Gouriet F, Oliver L, Jamme M, Casalta JP, Jimeno MT, Arregle F, Lavoute C, Hubert S, Philip M, Martel H, Riberi A, Habib G, Raoult D. High-dose trimethoprim-sulfamethoxazole and clindamycin for Staphylococcus aureus endocarditis. Int J Antimicrob Agents. 2019 Aug;54(2):143-148. doi: 10.1016/j.ijantimicag.2019.06.006. Epub 2019 Jun 8. PMID 31181351
- [Background] Suzuki J, Johnson J, Montgomery M, Hayden M, Price C. Outpatient Parenteral Antimicrobial Therapy Among People Who Inject Drugs: A Review of the Literature. Open Forum Infect Dis. 2018 Aug 7;5(9):ofy194. doi: 10.1093/ofid/ofy194. eCollection 2018 Sep. PMID 30211247
- [Background] Eaton EF, Mathews RE, Lane PS, Paddock CS, Rodriguez JM, Taylor BB, Saag MS, Kilgore ML, Lee RA. A 9-Point Risk Assessment for Patients Who Inject Drugs and Require Intravenous Antibiotics: Focusing Inpatient Resources on Patients at Greatest Risk of Ongoing Drug Use. Clin Infect Dis. 2019 Mar 5;68(6):1041-1043. doi: 10.1093/cid/ciy722. PMID 30165395
- [Background] Beieler AM, Dellit TH, Chan JD, Dhanireddy S, Enzian LK, Stone TJ, Dwyer-O'Connor E, Lynch JB. Successful implementation of outpatient parenteral antimicrobial therapy at a medical respite facility for homeless patients. J Hosp Med. 2016 Aug;11(8):531-5. doi: 10.1002/jhm.2597. Epub 2016 Apr 27. PMID 27120700
- [Background] Norris AH, Shrestha NK, Allison GM, Keller SC, Bhavan KP, Zurlo JJ, Hersh AL, Gorski LA, Bosso JA, Rathore MH, Arrieta A, Petrak RM, Shah A, Brown RB, Knight SL, Umscheid CA. 2018 Infectious Diseases Society of America Clinical Practice Guideline for the Management of Outpatient Parenteral Antimicrobial Therapy. Clin Infect Dis. 2019 Jan 1;68(1):e1-e35. doi: 10.1093/cid/ciy745. PMID 30423035
- [Background] Silverman M, Slater J, Jandoc R, Koivu S, Garg AX, Weir MA. Hydromorphone and the risk of infective endocarditis among people who inject drugs: a population-based, retrospective cohort study. Lancet Infect Dis. 2020 Apr;20(4):487-497. doi: 10.1016/S1473-3099(19)30705-4. Epub 2020 Jan 22. PMID 31981474
- [Background] Dagher M, Fowler VG Jr, Wright PW, Staub MB. A Narrative Review of Early Oral Stepdown Therapy for the Treatment of Uncomplicated Staphylococcus aureus Bacteremia: Yay or Nay? Open Forum Infect Dis. 2020 May 5;7(6):ofaa151. doi: 10.1093/ofid/ofaa151. eCollection 2020 Jun. PMID 32523971
- [Background] Tan C, Shojaei E, Wiener J, Shah M, Koivu S, Silverman M. Risk of New Bloodstream Infections and Mortality Among People Who Inject Drugs With Infective Endocarditis. JAMA Netw Open. 2020 Aug 3;3(8):e2012974. doi: 10.1001/jamanetworkopen.2020.12974. PMID 32785635
- [Background] Spellberg B, Chambers HF, Musher DM, Walsh TL, Bayer AS. Evaluation of a Paradigm Shift From Intravenous Antibiotics to Oral Step-Down Therapy for the Treatment of Infective Endocarditis: A Narrative Review. JAMA Intern Med. 2020 May 1;180(5):769-777. doi: 10.1001/jamainternmed.2020.0555. PMID 32227127